CLINICAL TRIAL: NCT03059862
Title: The Role of Tryptophan on Aryl Hydrocarbon Receptor Activation: a Randomized, Double Blind, Placebo-controlled, Crossover Design Pilot Trial
Brief Title: The Role of Dietary Tryptophan on Aryl Hydrocarbon Receptor Activation
Acronym: Aryl-IMMUNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: National Research Agency, France (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Aryl-IMMUNE
Record Dates: First submitted 2017-01-18; First posted 2017-02-23 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Diet Modification
Keywords: immunity; Aryl-hydrocarbon receptor; immune homeostasis; microbiota; tryptophan
MeSH Terms: interventions — Tryptophan

STUDY DESIGN:
Intervention Model Description: All subjects will be following a standardized low-tryptophan diet and randomized to L-tryptophan supplements or placebo, for three weeks. After a 2 weeks washout period, subjects will crossover to the other arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-tryptophan diet and L-tryptophan. (Experimental): Standardized low-tryptophan diet (500-1000 mg of L-tryptophan and 1800 kcal) + L-tryptophan supplements (3 g/day).
  Interventions: Dietary Supplement: L-tryptophan
- Low-tryptophan diet and placebo (Placebo Comparator): Standardized low-tryptophan diet (500-1000 mg of L-tryptophan and 1800 kcal) + placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-tryptophan — 3 g/day of L-tryptophan added to the standardized low-tryptophan diet. Duration: 3 weeks.
  Arms: Low-tryptophan diet and L-tryptophan.
Dietary Supplement: Placebo — A placebo will be added to the standardized low-tryptophan diet. Duration: 3 weeks.
  Arms: Low-tryptophan diet and placebo

SUMMARY:
This study evaluates the role of dietary L-tryptophan, an essential amino acid, in the activation of a specific cellular component: the aryl hydrocarbon receptor.

DETAILED DESCRIPTION:
The Aryl hydrocarbon receptor (AHR) is a ligand-dependent transcription factor implicated in a range of key cellular events. In the gut, AHR is crucial for maintaining intestinal barrier immune homeostasis. The physiology of the AHR, however, is not completely understood; its precise gut luminal activators and functional consequences are unknown.

Some AHR ligands originate from the diet. Commensals play crucial roles in metabolizing tryptophan and other amino acids such as tyrosine, with the subsequent production of tryptophan metabolites. Previous studies show that inflammatory bowel disease (IBD) patients have impaired production of AHR agonists by the microbiota. Furthermore, dietary supplementation with tryptophan ameliorates clinical parameters of colitis in rodent models. Whether these findings translate into human pathophysiology has not been explored.

In the present study, the investigators will evaluate the effect of high- versus low-tryptophan diet on AHR activation in healthy participants. Briefly, participants will be instructed to follow a standardized low-tryptophan diet and will be randomized to a 3-week L-tryptophan supplement or placebo. Later, after a 2-week washout period, participants will crossover to the other arm. In addition, the effect of tryptophan and microbiota-derived metabolites on AHR activation will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between 18 and 75 years of age.

Exclusion Criteria:

* Rome IV criteria for any functional gastrointestinal disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
AHR activation levels in stool and duodenal content. | three weeks
  Changes in AHR activation levels will be assessed in stool and duodenal samples before and after the intervention (high- and low-tryptophan diets) using an AHR cell-reporter line.

SECONDARY OUTCOMES:
Bacterial and fungal microbiota composition in stool, duodenum and rectum/sigmoid biopsies. | Three weeks
  Changes in bacterial and fungal microbiota composition will be assessed before and after the intervention in stool samples, duodenum and rectum biopsies.
Tryptophan metabolites levels, including host and bacterial catabolites, in blood, urine and stool. | Three weeks
  Changes in tryptophan metabolites leves will be compared before and after the intervention, in blood, urine and stool samples.
mRNA levels in duodenal and rectum/sigmoid biopsies. | three weeks
  Changes in mRNA levels in duodenal and rectum/sigmoid biopsies will be assessed before and after the intervention.
Cytokines in serum. | three weeks.
  Changes in cytokines in the serum (IL-22, IL-6, IL-2, IL-10, IL-12p70, IL-23p19, IFNγ, TNFα and CRP will be measured by ELISA in cell culture supernatants after stimulation with LPS, curdlan and ConA ) will be measured before and after the intervention and patients will be grouped into two categories for each measurement: high vs. low, according to the cutoff reference test value for each of the cytokines.
Gastrointestinal symptoms | three weeks.
  Changes in gastrointestinal symptoms before and after the intervention will be assessed using a validated questionnaire (The Gastrointestinal Symptoms Rating Scale)
Mood | three weeks
  Changes in mood before and after the intervention will be assessed using a validated questionnaire (Hospital anxiety and depression scale)

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Bercik, MD, PhD, Principal Investigator — McMaster University, Department of Medicine, Division of Gastroenterology
Locations (1):
- McMaster Health Sciences Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barouki R, Coumoul X, Fernandez-Salguero PM. The aryl hydrocarbon receptor, more than a xenobiotic-interacting protein. FEBS Lett. 2007 Jul 31;581(19):3608-15. doi: 10.1016/j.febslet.2007.03.046. Epub 2007 Mar 30. PMID 17412325
- [Background] Behnsen J, Raffatellu M. Keeping the peace: aryl hydrocarbon receptor signaling modulates the mucosal microbiota. Immunity. 2013 Aug 22;39(2):206-7. doi: 10.1016/j.immuni.2013.08.012. PMID 23973218
- [Background] Bender DA. Biochemistry of tryptophan in health and disease. Mol Aspects Med. 1983;6(2):101-97. doi: 10.1016/0098-2997(83)90005-5. No abstract available. PMID 6371429
- [Background] Cynober L, Bier DM, Kadowaki M, Morris SM Jr, Elango R, Smriga M. Proposals for Upper Limits of Safe Intake for Arginine and Tryptophan in Young Adults and an Upper Limit of Safe Intake for Leucine in the Elderly. J Nutr. 2016 Dec;146(12):2652S-2654S. doi: 10.3945/jn.115.228478. Epub 2016 Nov 9. PMID 27934658
- [Background] Hubbard TD, Murray IA, Bisson WH, Lahoti TS, Gowda K, Amin SG, Patterson AD, Perdew GH. Adaptation of the human aryl hydrocarbon receptor to sense microbiota-derived indoles. Sci Rep. 2015 Aug 3;5:12689. doi: 10.1038/srep12689. PMID 26235394
- [Background] Kiss EA, Vonarbourg C, Kopfmann S, Hobeika E, Finke D, Esser C, Diefenbach A. Natural aryl hydrocarbon receptor ligands control organogenesis of intestinal lymphoid follicles. Science. 2011 Dec 16;334(6062):1561-5. doi: 10.1126/science.1214914. Epub 2011 Oct 27. PMID 22033518
- [Background] Kiss EA, Vonarbourg C. Aryl hydrocarbon receptor: a molecular link between postnatal lymphoid follicle formation and diet. Gut Microbes. 2012 Nov-Dec;3(6):577-82. doi: 10.4161/gmic.21865. Epub 2012 Aug 22. PMID 22909905
- [Background] Li Y, Innocentin S, Withers DR, Roberts NA, Gallagher AR, Grigorieva EF, Wilhelm C, Veldhoen M. Exogenous stimuli maintain intraepithelial lymphocytes via aryl hydrocarbon receptor activation. Cell. 2011 Oct 28;147(3):629-40. doi: 10.1016/j.cell.2011.09.025. Epub 2011 Oct 13. PMID 21999944
- [Background] Zelante T, Iannitti RG, Cunha C, De Luca A, Giovannini G, Pieraccini G, Zecchi R, D'Angelo C, Massi-Benedetti C, Fallarino F, Carvalho A, Puccetti P, Romani L. Tryptophan catabolites from microbiota engage aryl hydrocarbon receptor and balance mucosal reactivity via interleukin-22. Immunity. 2013 Aug 22;39(2):372-85. doi: 10.1016/j.immuni.2013.08.003. PMID 23973224
- [Background] Qiu J, Heller JJ, Guo X, Chen ZM, Fish K, Fu YX, Zhou L. The aryl hydrocarbon receptor regulates gut immunity through modulation of innate lymphoid cells. Immunity. 2012 Jan 27;36(1):92-104. doi: 10.1016/j.immuni.2011.11.011. Epub 2011 Dec 15. PMID 22177117
- [Result] Lamas B, Richard ML, Leducq V, Pham HP, Michel ML, Da Costa G, Bridonneau C, Jegou S, Hoffmann TW, Natividad JM, Brot L, Taleb S, Couturier-Maillard A, Nion-Larmurier I, Merabtene F, Seksik P, Bourrier A, Cosnes J, Ryffel B, Beaugerie L, Launay JM, Langella P, Xavier RJ, Sokol H. CARD9 impacts colitis by altering gut microbiota metabolism of tryptophan into aryl hydrocarbon receptor ligands. Nat Med. 2016 Jun;22(6):598-605. doi: 10.1038/nm.4102. Epub 2016 May 9. PMID 27158904